CLINICAL TRIAL: NCT03482440
Title: Role of Angiotensin II and Chronic Inflammation in Persistent Microvascular Dysfunction Following Preeclamptic Pregnancy
Brief Title: Angiotensin II and Chronic Inflammation in Persistent Microvascular Dysfunction Following Preeclampsia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: Penn State University (Other)
Responsible Party: Principal Investigator, Anna Stanhewicz, PhD, Principal Investigator, University of Iowa
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 201909818
Record Dates: First submitted 2018-03-15; First posted 2018-03-29 (Actual); Results first posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Preeclampsia
Keywords: preeclampsia; microvascular; inflammation; angiotensin II
MeSH Terms: conditions — Pre-Eclampsia; Inflammation | interventions — salicylsalicylic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet
- Salsalate (Experimental)
  Interventions: Drug: Salsalate Oral Tablet

INTERVENTIONS:
Drug: Salsalate Oral Tablet — 1500mg twice daily for 4 days prior to experimental testing
  Arms: Salsalate
Drug: Placebo Oral Tablet — Placebo oral table twice daily for 4 days prior to experimental testing
  Arms: Placebo

SUMMARY:
Women who develop preeclampsia during pregnancy are more likely to develop cardiovascular disease later in life, even if they are otherwise healthy. The reason why this occurs is unclear but may be related to blood vessel damage and increased inflammation that occurs during the preeclamptic pregnancy and persists postpartum. The purpose of this investigation is to 1) determine the mechanisms contributing to this lasting blood vessel damage and chronic inflammation, and to 2) identify factors (both physiological and pharmacological) that mitigate these negative effects in order to inform better clinical management of cardiovascular disease risk in women who have had preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Post-partum women who have delivered within two years and who have had a preeclamptic pregnancy diagnosed by their obstetrician before 34 weeks of gestation and confirmed according to the American College of Obstetricians and Gynecologists criteria for severe preeclampsia. [This information will be self-reported by the subjects.]
* Post-partum women who have delivered within two years and who have had a normal pregnancy.
* 18 years and older.

Exclusion Criteria:

* skin diseases
* current tobacco use
* diagnosed or suspected hepatic or metabolic disease
* statin or other cholesterol-lowering medication
* history of hypertension prior to pregnancy
* history of gestational diabetes
* current pregnancy
* allergy to aspirin or NSAIDs or known allergy to materials used during the experiment (e.g. latex)
* renal disease, bleeding disorders and history of gastrointestinal bleeding.
* Known allergies to study drugs
* Taking blood thinners, aspirin or NSAIDS.
* Women who choose to breastfeed will not participate in any parts of the project that include salsalate.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-08-26 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Stanhewicz, PhD, Principal Investigator — University of Iowa
Locations (2):
- United States (2):
  - University of Iowa, Iowa City, Iowa
  - Pennsylvania State University, University Park, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: this is a crossover study design - all participants (23 total) completed each arm of the study in a randomized placebo controlled study design
Groups:
- Placebo Then Salsalate: Placebo oral table twice daily for 4 days prior to experimental testing followed by 14 day washout period and then salsalate oral tablet 1500mg twice daily for 4 days prior to experimental testing
- Salsalate Then Placebo: Salsalate Oral Tablet 1500mg twice daily for 4 days prior to experimental testing followed by 14 day washout period and then placebo oral tablet twice daily for 4 days prior to experimental testing
Period: Overall Study
Arm/Group | Placebo Then Salsalate | Salsalate Then Placebo
Started | 13 | 10
Completed | 13 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All participants were randomized to received both interventions.
Arm/Group | All Study Participants
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Microvascular Endothelial Function (Cutaneous Conductance, %Maximum)
Description: Endothelium-dependent vasodilation assessed as cutaneous conductance response (cutaneous conductance = local red blood cell flux/mean arterial pressure; %maximum) to exogenous acetylcholine delivered via intradermal microdialysis.
Time Frame: immediately following the 4 days or oral treatment (salsalate or placebo)
Measure: Mean (Standard Deviation); unit: % of maximal cutaneous conductance
Groups:
- Oral Salsalate: Participants first received 4 days oral salsalate tablet 1500mg twice daily.
- Oral Placebo: Participants first received 4 days of placebo treatment twice daily.
Arm/Group | Oral Salsalate | Oral Placebo
Number analyzed (Participants) | 23 | 23
% of maximal cutaneous conductance | 95 (6) | 77 (8)

2. Secondary Outcome: Peripheral Blood Mononuclear Cell Inflammatory Response to Ang II
Description: inflammatory cytokine (TNFalpha) release by peripheral blood mononuclear cells isolated from fresh whole blood collected via venipuncture and stimulated with angiotensin II ex vivo.
Time Frame: at the completion of 4 days of oral (placebo or salsalate) treatment
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Oral Salsalate: Participants who received 4 days oral salsalate tablet 1500mg twice daily.
- Oral Placebo: Participants who received 4 days oral placebo tablet.
Arm/Group | Oral Salsalate | Oral Placebo
Number analyzed (Participants) | 23 | 23
ng/ml | 2.37 (1.28) | 2.77 (1.01)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected on day 2 and day 4 of the 4 day treatment periods.
Groups:
- Placebo: Placebo oral table twice daily for 4 days prior to experimental testing.
- Salsalate: Salsalate Oral Tablet 1500mg twice daily for 4 days prior to experimental testing.
Arm/Group | Placebo | Salsalate
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 2/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=23) | Salsalate (N=23)
tennitis while on salsalate (Ear and labyrinth disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/40/NCT03482440/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-24): https://cdn.clinicaltrials.gov/large-docs/40/NCT03482440/ICF_001.pdf